CLINICAL TRIAL: NCT06220669
Title: An Adaptive Phase 2a/2b, Randomized, Double-Blind, Parallel-Group Study to Investigate the Safety and Efficacy of LY3541860 Compared to Placebo in Slowing the Occurrence of New T1 Gadolinium-Enhancing Lesions in Adult Participants With Relapsing Multiple Sclerosis
Brief Title: A Study of LY3541860 in Adult Participants With Relapsing Multiple Sclerosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18548; J3K-MC-KIAB (Other: Eli Lilly and Company); 2023-503289-22-00 (Other: EU Trial Number)
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing remitting multiple sclerosis, Clinically isolated syndrome, Secondary progressive multiple sclerosis with disease activity.
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- LY3541860 Phase 2a Dose Level 1 (Experimental): LY3541860 will be given intravenously (IV)
  Interventions: Drug: LY3541860
- LY3541860 Phase 2a Dose Level 2 (Experimental): LY3541860 will be given IV.
  Interventions: Drug: LY3541860
- Placebo Phase 2a (Placebo Comparator): Placebo will be given IV.
  Interventions: Drug: Placebo
- LY3541860 Phase 2b Dose Level 3 (Experimental): LY3541860 will be given IV.
  Interventions: Drug: LY3541860
- LY3541860 Phase 2b Dose Level 4 (Experimental): LY3541860 will be given IV.
  Interventions: Drug: LY3541860
- Placebo Phase 2b (Placebo Comparator): Placebo will be given IV.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3541860 — Administered IV
  Arms: LY3541860 Phase 2a Dose Level 1; LY3541860 Phase 2a Dose Level 2; LY3541860 Phase 2b Dose Level 3; LY3541860 Phase 2b Dose Level 4
Drug: Placebo — Administered IV
  Arms: Placebo Phase 2a; Placebo Phase 2b

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of LY3541860 in adult participants with multiple sclerosis that gets worse and gets better. The study will last about 9 months with additional 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet criteria for relapsing forms of multiple sclerosis, including relapsing-remitting multiple sclerosis based on the 2017 revision of the McDonald diagnostic criteria (Thompson et al. 2018) with a relapsing course (RMS) activity according to Klineova and Lublin 2018.
* Participants must have 1 of these:

  * at least 1 documented relapse within the previous year
  * at least 2 documented relapses within the previous 2 years, or
  * at least 1 active GdE brain lesion on an MRI scan in the past 180 days prior to screening.
* Have an Expanded Disability Status Scale (EDSS) score of less than or equal to (≤) 5.5 at screening and randomization.

Exclusion Criteria:

* Have had a diagnosis of:

  * primary progressive multiple sclerosis (MS) according to the 2017 revision of McDonald diagnostic criteria (Thompson et al. 2018), or
  * nonactive secondary progressive MS ( Klineova and Lublin 2018).
* Meet criteria for neuromyelitis optica spectrum disorder (Wingerchuk and Lucchinetti 2022).
* Have a history of clinically significant central nervous system (CNS) disease.
* Have had a confirmed relapse with systemic corticosteroid administration <30 days prior to randomization.
* Have more than 20 active GdE brain lesions on screening MRI scan.
* Have received any of these medications or treatments.
* Have a current or recent acute, active infection.
* Have current serious or unstable illnesses.
* Have any other clinically important abnormality at screening or baseline.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Cumulative Number of New T1 Gadolinium-Enhancing (GdE) Lesions | 12 Weeks
  Cumulative number will be measured by magnetic resonance imaging (MRI) scans.

SECONDARY OUTCOMES:
Cumulative Number of Total Number of T1 GdE Lesions | 12 Weeks
  Cumulative number will be measured by MRI scans.
Cumulative Number of New and/or Enlarging T2 Lesions | 12 Weeks
  Cumulative number will be measured by MRI scans.
Pharmacokinetics (PK): Plasma Trough Concentrations of LY3541860 | Baseline Through Week 12
  Plasma trough concentrations of LY3541860 was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (50):
- United States (16):
  - Healthcare Innovations Institute, LLC, Coral Springs, Florida
  - Royal Palm Medical Group, Fort Myers, Florida
  - Eastern Medical Group Research, Fort Myers, Florida
  - Panhandle Research and Medical Clinic, Gulf Breeze, Florida
  - High Quality Research, Miami, Florida
  - USF MS Center, Tampa, Florida
  - Conquest Research LLC - Winter Park - ClinEdge - PPDS, Winter Park, Florida
  - Consultants in Neurology, Northbrook, Illinois
  - Sharlin Health and Neurology, Ozark, Missouri
  - Psych Care Consultants Research, St Louis, Missouri
  - Premier Neurology, Greer, South Carolina
  - Hope Neurology, Knoxville, Tennessee
  - ANRC Research, El Paso, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - 1960 Family Practice, PA, Houston, Texas
  - Swedish Multiple Sclerosis Center, Seattle, Washington
- France (4):
  - Centre Hospitalier Universitaire de Clermont Ferrand, Clermont-Ferrand
  - CHRU de Nancy, Nancy
  - CHU Gui De Chauliac, Nîmes
  - Centre Hospitalier Intercommunal - Site de Poissy, Poissy
- Germany (8):
  - Zentrum für klinische Forschung Dr. med. Irma Schöll, Bad Homburg
  - Klinikum Bayreuth GmbH, Bayreuth
  - Studienzentrum für Neurologie und Psychiatrie, Böblingen
  - Universitatsklinikum Leipzig, Leipzig
  - Institut für klinische Neuroimmunologie LMU Muenchen, München
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen
  - Nervenfachärztliche Gemeinschaftspraxis Ulm, Ulm
- Israel (2):
  - Galilee Medical Center, Nahariya
  - Kaplan Medical Center, Rehovot
- Italy (3):
  - Fondazione Istituto G. Giglio di Cefalù, Cefalù
  - Ospedale San Raffaele S.r.l. - PPDS, Milan
  - Fondazione IRCCS Di Rilievo Nazionale Istituto Nazionale Neurologico Carlo Besta-VIA MANGIAGALLI 3, Milan
- Pauls Stradins Clinical Univeristy Hospital, Riga, Latvia
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda Hospital, Affiliate of Klaipeda University Hospital, Klaipėda
- Poland (12):
  - Neurocentrum Bydgoszcz sp. z o.o., Bydgoszcz
  - Specjalistyczna Praktyka Lekarska prof. Grzegorz Opala, Katowice
  - M.A. - LEK A.M. Maciejowscy SC. Centrum Terapii SM, Katowice
  - NEURO-MEDIC Sp. z o. o., Katowice
  - Clinirem, Lublin
  - Med-Polonia Sp. z o.o., Poznan
  - Niepubliczny Zaklad Opieki Zdrowotnej NEURO-KARD Ilkowski i Partnerzy Spolka Partnerska Lekarzy, Poznan
  - Centrum Medyczne NeuroProtect, Warsaw
  - ETG Neuroscience - PPDS, Warsaw
  - Neurosphera SP. Z O.O, Warsaw
  - IBISMED Wielospecjalistyczne Centrum Medyczne, Zabrze
  - ProNeuro Centrum Medyczne, Żory
- Nemocnica Ruzinov, Bratislava, Slovakia
- Queen's Medical Centre, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/453415